CLINICAL TRIAL: NCT07128030
Title: Moderate-Intensity Exercise and Pain Sensitization in Breast Cancer Survivors: A Case-Based Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, DeAsís-Fernández, Francisco, Director, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EDCM
Record Dates: First submitted 2025-07-25; First posted 2025-08-17 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Exercise Training; Breast Cancer; Pain Management
Keywords: pain severity; pain sensibilization; quantitative sensory testing; physical activity
MeSH Terms: conditions — Breast Neoplasms; Agnosia; Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Intensity Exercise (Experimental): The experimental group followed a structured five-week program combining moderate-intensity aerobic and resistance training, totaling 150 minutes per week, and supervised by physiotherapists. Exercise intensity was monitored using the Borg and OMNI-Res perceived exertion scales, with prior familiarization sessions provided. Adherence was supported through attendance tracking, reminder messages, and motivational feedback. Unlike previous studies focused on fatigue or quality of life, this protocol targeted pain modulation based on neurophysiological mechanisms. Sessions included step-based aerobic routines and resistance exercises with bands, with clear safety and effort guidelines in place. No drugs or devices were used during the intervention.
  Interventions: Other: Exercise
- Control Group (No Intervention): Participants maintained usual activities for five weeks without changing exercise habits. No additional interventions (drugs, devices, or procedures) were applied.

INTERVENTIONS:
Other: Exercise — The experimental group completed a five-week supervised program combining moderate-intensity aerobic and resistance training (150 min/week). Intensity was monitored using the Borg and OMNI-Res scales after familiarization sessions. Adherence was encouraged through reminders, motivational messages, and follow-ups. Unlike prior studies, this intervention focused specifically on neurophysiological pain modulation. Sessions included step-based aerobic exercises and resistance training with elastic bands under safety protocols.
  Arms: Moderate-Intensity Exercise

SUMMARY:
The aim of this study was to evaluate the feasibility, safety, and acceptability of a supervised, combined moderate-intensity aerobic and resistance training program designed to reduce pain sensitization in BCS with persistent pain. Secondary objectives included assessing changes in pain intensity, somatosensory sensitivity, and temporal summation, while tertiary objectives focused on improvements in quality of life and functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Adult women diagnosed with stage I-III breast cancer
* Completion of active treatment (surgery, chemotherapy, and/or radiotherapy) at least 6 months prior to enrollment
* Presence of persistent pain or altered sensation in the upper quadrant of the affected limb related to oncologic treatment

Exclusion Criteria:

* Bilateral breast cancer
* Locoregional recurrence
* Other malignancies
* Pre-existing pain not related to cancer treatment
* Neurological or cognitive disorders
* Non-Spanish speakers
* Contraindications to moderate-intensity physical activity

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2025-08-23 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Adherence by Tolerance: number of incomplete sessions | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  This variable captures tolerance-related indicators, including number of incomplete sessions. This variable will be analyzed using contingency tables to evaluate therapeutic adherence based on tolerance.
Adherence by Tolerance: number of sessions at moderate intensity | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  This variable captures tolerance-related indicators, including number of sessions at moderate intensity. This variable will be analyzed using contingency tables to evaluate therapeutic adherence based on tolerance.
Adherence by Tolerance: number of participants completing at moderate intensity | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  This variable captures tolerance-related indicators, including number of participants completing at moderate intensity. This variable will be analyzed using contingency tables to evaluate therapeutic adherence based on tolerance.
Adherence by Tolerance: number of progressions during the program | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  This variable captures tolerance-related indicators, including number of progressions during the program. This variable will be analyzed using contingency tables to evaluate therapeutic adherence based on tolerance.
Adherence by Tolerance: final progression level reached | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  This variable captures tolerance-related indicators, including final progression level reached. This variable will be analyzed using contingency tables to evaluate therapeutic adherence based on tolerance.
Adherence by Motivation: number of absences | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  This variable aggregates motivation-related indicators, including number of absences.This variable will be analyzed using contingency tables to evaluate therapeutic adherence based on motivation.
Adherence by Motivation: percentage of sessions recovered after absence | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  This variable aggregates motivation-related indicators, including percentage of sessions recovered after absence. This variable will be analyzed using contingency tables to evaluate therapeutic adherence based on motivation.
Adherence by Motivation: number of dropouts | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  This variable aggregates motivation-related indicators, including number of dropouts.This variable will be analyzed using contingency tables to evaluate therapeutic adherence based on motivation.
Adherence by Motivation: number of presence of positive sensations | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  This variable aggregates motivation-related indicators, including number of presence of positive sensations (e.g., satisfaction, motivation).This variable will be analyzed using contingency tables to evaluate therapeutic adherence based on motivation.
Adherence by Motivation: number of occurrence of adverse effects | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  This variable aggregates motivation-related indicators, including number of occurrence of adverse effects.This variable will be analyzed using contingency tables to evaluate therapeutic adherence based on motivation.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  The BPI consists of 11 items: four assessing intensity and seven evaluating interference in areas such as general activity, mood, walking ability, work, relationships, sleep, and enjoyment of life. Scores range from 0 to 10, with higher scores indicating greater pain or interference. The BPI has demonstrated strong test-retest reliability (0.59-0.94), internal consistency in cancer populations (Cronbach's alpha 0.81-0.89), and construct validity across various demographic and clinical subgroups
Numerical Rating Scale (NRS) | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  Pain intensity was measured using the Numerical Rating Scale (NRS), which ranges from 0 ("no pain") to 10 ("worst imaginable pain"). This scale has shown high reproducibility in assessing pain exacerbations (Cohen's κ = 0.86) and overall pain intensity (Cohen's κ = 0.80)
Self-report Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  A validated Spanish-language tool composed of seven yes/no items, with scores ranging from 0 to 24. A score of 12 or higher indicates a high probability of neuropathic pain, while a score below 12 suggests a low likelihood. The S-LANSS has demonstrated strong diagnostic properties, with 85% sensitivity and 80% specificity
SENSORIMOTOR CHARACTERISTICS: HANDGRIP STRENGTH | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  Handgrip strength was assessed using a Jamar hydraulic dynamometer set to the second handle position. Participants performed three 5-second maximal isometric contractions per hand, with 30-second rests between attempts. The average of the three trials was used for analysis, starting with the non-operated side. Standardized verbal instructions and countdowns were given to ensure consistency.
Somatosensorial status (QST): MECHANICAL DETECTION THRESHOLD (MDT) | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  Calibrated Von Frey monofilaments were applied perpendicularly to the skin until the filament just bent. Filament sizes were increased until the first sensation was detected, and the initial detectable filament was recorded. A descending series was then applied to identify the smallest filament still perceived. This ascending-descending method was repeated five times, and the method of limits was used to determine thresholds.
  Standardized instructions: "With your eyes open, I will apply pressure using several filaments of varying stiffness. Some you may feel, others you may not. Then, with your eyes closed, please indicate each time you feel the stimulus. Close your eyes, and we will begin."
Somatosensorial status (QST): MECHANICAL PAIN THRESHOLD (MPT) | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  Mechanical pain threshold was assessed using Von Frey filaments. Filaments were applied in ascending order until the participant first reported the sensation as painful. Then, a descending sequence identified the smallest filament still perceived as painful. The test was repeated five times, and the mean filament force (measured in grams) was recorded as the MPT.
  Standardized instructions: "You will feel a sharp stimulus. Please tell me when the sensation becomes uncomfortable but not yet painful-approximately 4 out of 10 on the Numerical Pain Rating Scale (NPRS), where 0 = no pain and 10 = worst imaginable pain. Higher filament force indicates a higher pain threshold (less sensitivity)."
Somatosensorial status (QST): PAIN FACILITATION | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  Temporal summation was evaluated using Von Frey filaments at the mechanical pain threshold. A single stimulus was applied to a fixed point, followed by a pain rating on the NRS (, 0-10). Then, 10 identical stimuli were delivered at a frequency of 1 Hz using a 60- bpm metronome. A second NRS score was collected immediately after. The procedure was repeated three times, and the average was used for analysis.
  Standardized instructions: "We will apply the same sharp stimulus used in the previous test. Please rate your pain intensity on a scale from 0 to 10, where 0 means no pain and 10 indicates the worst imaginable pain. Keep your eyes closed during the procedure. First, rate your pain after one stimulus, and then again after the sequence of ten."
Somatosensorial status (QST): PRESSURE PAIN THRESHOLD (PPT) | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  Pressure pain threshold was measured using a digital algometer (Wagner Instruments FPX 100). With the patient in a supine position, incremental pressure was applied perpendicularly to the skin until pain was first perceived. Three measurements were obtained per site, and the average was used for analysis. Assessments were conducted at the primary painful area, the contralateral upper limb, and the anterior thigh of a pain-free lower limb.
Physical activity was assessed using the Global Physical Activity Questionnaire (GPAQ) | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  A self-reported instrument developed by the World Health Organization and validated for use in cancer populations and Spanish-speaking individuals. The GPAQ evaluates physical activity in three domains-occupational, transportation, and leisure-and also captures sedentary behavior, defined as daily time spent sitting or lying down, excluding sleep. Based on total activity scores, participants were classified as inactive (<100), mildly active (100-1951), moderately active (1952-5724), or vigorously active (≥5725) (Cleland et al., 2014).
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Breast Cancer Module (EORTC QLQ-BR23). | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  This 23-item questionnaire includes four functional scales (body image, sexual functioning, sexual enjoyment, and future perspective) and four symptom scales (side effects of therapy, breast symptoms, arm symptoms, and distress from hair loss). Responses are given on a 4-point Likert scale ranging from 0 ("not at all") to 4 ("very much")
CARDIOPULMONARY FITNESS | Baseline (prior to intervention), immediately post-intervention (within 1 week), and at 6-month follow-up.
  Functional capacity was assessed using the Siconolfi Step Test, a validated submaximal test for estimating maximal oxygen uptake (VO₂max) in cancer populations. The test was performed on a 10-inch (25.4 cm) step in three 3-minute stages, with 1-minute rest intervals. Cadence was controlled via metronome at 68 bpm (stage 1), 104 bpm (stage 2), and 136 bpm (stage 3), corresponding to 17, 26, and 32 steps per minute, respectively. Heart rate was recorded at 2:30 minutes into each stage using a POLAR monitor. The test was terminated if participants experienced cardiorespiratory symptoms, musculoskeletal discomfort, peripheral fatigue, inability to maintain cadence, an RPE of 10, or if heart rate exceeded 65% of age-predicted maximum (220 - age).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No